CLINICAL TRIAL: NCT02692170
Title: A Single Center, Randomized, Double Blinded PhaseI/IIa Exploratory Study to Evaluate Reactogenicity, Safety, Immunogenicity and Dose Response of a New Hepatitis B Vaccine in Human Adult
Brief Title: A Study to Evaluate the Reactogenicity, Safety, and Immunogenicity of the Third Generation Hepatitis B Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHA Vaccine Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CVI-HBV-001-CT1201
Record Dates: First submitted 2016-02-18; First posted 2016-02-25 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CVI-HBV-001 (5 μg) (Experimental): * HBV surface antigen 5 μg/dose
  * Intramuscular injection at 0, 1, 6th month
  Interventions: Biological: CVI-HBV-001
- CVI-HBV-001 (10 μg) (Experimental): * HBV surface antigen 10 μg/dose
  * Intramuscular injection at 0, 1, 6th month
  Interventions: Biological: CVI-HBV-001
- CVI-HBV-001 (20 μg) (Experimental): * HBV surface antigen 20 μg/dose
  * Intramuscular injection at 0, 1, 6th month
  Interventions: Biological: CVI-HBV-001
- CVI-HBV-001 (40 μg) (Experimental): * HBV surface antigen 40 μg/dose
  * Intramuscular injection at 0, 1, 6th month
  Interventions: Biological: CVI-HBV-001
- Conventional Hepatitis B vaccine (20 μg) (Active Comparator): * HBV surface antigen 20 μg/dose
  * Intramuscular injection at 0, 1, 6th month
  Interventions: Biological: Conventional Hepatitis B vaccine (20 μg)

INTERVENTIONS:
Biological: CVI-HBV-001 — Investigational Product
  Arms: CVI-HBV-001 (10 μg); CVI-HBV-001 (20 μg); CVI-HBV-001 (40 μg); CVI-HBV-001 (5 μg)
Biological: Conventional Hepatitis B vaccine (20 μg) — Investigational Product
  Arms: Conventional Hepatitis B vaccine (20 μg)

SUMMARY:
A single center, randomized, double blinded phase I/IIa exploratory study to evaluate reactogenicity, safety, immunogenicity and dose-response of a new hepatitis B vaccine in human adult

DETAILED DESCRIPTION:
* Objectives: To explore the most effective dose of the third generation Hepatitis B vaccine through the evaluation of reactogenicity, safety, and immunogenicity.
* Subjects: Adults having anti-HBs antibody titers less than 10 mIU/mL after 3 previous injections of the conventional Hepatitis B vaccine.
* Study hypothesis: The third generation Hepatitis B vaccine, containing preS antigens in addition to S antigen, has an ability to elicit faster protection and higher antibody titers than the second generation Hepatitis B vaccine in the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 20 and 50 years of age
2. Anti-HBs titers < 10 mIU/mL
3. Subject is able to provide written informed consent by oneself or legal representative

Exclusion Criteria:

1. Hepatitis B core antibodies positive patient
2. Patient has abnormal results in liver-function test
3. Patient has active microbial, viral, or fungal infections in need of systemic treatment
4. Patient has history of serious heart disease (NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, treatment required ventricular tachyarrhythmias, or unstable angina etc.)
5. Patient has seizure disorder required anticonvulsants treatment
6. Serious chronic obstructive pulmonary disease patient accompanied hypoxemia
7. Uncontrollable diabetic patient
8. Uncontrollable hypertension patient
9. Patient with known history of HIV, HBV, or HCV infection
10. Subject had experience of participating other clinical study or clinical treatment within 30 days before screening
11. Subject has hypersensitivity or anaphylactic reaction for HBV vaccine components
12. Patient being treated for prolonged immunosuppressive therapy (including steroids)
13. Hemodialysis patient
14. Subject has continuous drinking (>21 units/week, 1 unit = 10g of pure alcohol) or dependence on alcohol
15. Subject is pregnant or breastfeeding or intending to become pregnant during the study
16. Subject has any other significant findings unacceptable in this study under the opinion of the investigator

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2015-05-28 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity (including incidence of adverse events and expected adverse reactions for vaccine treatment) measured for 7 days after each vaccination | 7 days after each vaccination
  Occurrence of severe local and/or systemic reactogenicity signs and symptoms measured for 7 days after each vaccination

SECONDARY OUTCOMES:
Seroprotection rate | 4 weeks after vaccination
  Seroprotection (> 10 mIU/mL of anti-HBs) rate measured 4 weeks after vaccination
Antibody titers to HBsAg | 4 weeks after vaccination
  Geometric mean titer (GMT, mIU/mL) measured 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Seong Gyu Hwang, M.D., Ph.D., Principal Investigator — Bundang CHA General Hospital